CLINICAL TRIAL: NCT00544011
Title: Phase II Study Evaluating the Association of Bevacizumab and Chemotherapy of the Type Modified FOLFIRI 3 in Patients With Metastatic Colorectal Adenocarcinoma
Brief Title: Bevacizumab and Combination Chemotherapy in Treating Patients With Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hopital Jean Minjoz (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Purpose: Treatment
Other Study IDs: CDR0000564118; CHRB-Folfiri-III-Avastin; INCA-RECF0432
Record Dates: First submitted 2007-10-13; First posted 2007-10-16 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2009-07

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Bevacizumab; Capecitabine; Fluorouracil; Irinotecan

INTERVENTIONS:
Biological: bevacizumab
Drug: capecitabine
Drug: fluorouracil
Drug: irinotecan hydrochloride
Other: diagnostic laboratory biomarker analysis

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Drugs used in chemotherapy, such as irinotecan, fluorouracil, and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving bevacizumab together with combination chemotherapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well bevacizumab given together with combination chemotherapy works in treating patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the objective response (complete and partial) rate in patients with metastatic colorectal adenocarcinoma treated with bevacizumab and modified FOLFIRI 3 chemotherapy.

Secondary

* Determine progression-free and overall survival.
* Determine the tolerance to this regimen.
* Evaluate the resectability rate.
* Evaluate biological markers predictive of the efficacy of this regimen.

OUTLINE: This is a multicenter study.

Patients receive bevacizumab IV over 30-90 minutes on day 1, irinotecan hydrochloride IV over 90 minutes on days 1 and 3, and fluorouracil IV continuously over 46 hours on day 1. Treatment repeats every 2 weeks for up to 12 courses in the absence of disease progression or unacceptable toxicity.

At 14 days after completing chemotherapy, patients with progressive or stable disease receive maintenance therapy comprising bevacizumab and capecitabine.

Biological specimens are collected at baseline and before the fourth course of chemotherapy.

After completion of study therapy, patients are followed every 3 months for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the colon or rectum

  * Previously untreated metastatic disease
* Measurable disease by RECIST

  * Must not be located in a prior radiation field
* No cerebral or meningeal metastases

PATIENT CHARACTERISTICS:

Inclusion criteria:

* WHO performance status 0-1
* Life expectancy > 12 weeks
* Absolute neutrophil count ≥ 1,000/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Transaminases ≤ 2 times ULN (5 times ULN if liver metastases present)
* Alkaline phosphatase ≤ 2 times ULN (5 times ULN if liver metastases present)
* Creatinine ≤ 130 μmol/L OR creatinine clearance ≥ 30 mL/min
* Proteinuria < 2+ or urine protein ≤ 1 g/24 hours
* Not pregnant or nursing
* Fertile patients of must use effective contraception

Exclusion criteria:

* Uncontrolled cardiac disease
* Prior cerebral vascular accident
* Uncontrolled arterial hypertension
* Severe renal or hepatic insufficiency
* Prior arteriopathy
* Bleeding disorder or nonhealing wound
* Coagulopathy
* Other malignancy within the past 2 years except basal cell or squamous cell skin cancer or curatively treated carcinoma of the cervix
* Psychiatric disorder compromising comprehension or participation in the study
* Intestinal occlusion or subocclusion not caused by medical therapy

PRIOR CONCURRENT THERAPY:

Inclusion criteria:

* See Disease Characteristics

Exclusion criteria:

* Prior adjuvant bevacizumab or irinotecan hydrochloride
* Concurrent aspirin (> 325 mg/day) or therapeutic anticoagulants
* Surgery in the past 28 days

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2007-04

PRIMARY OUTCOMES:
Objective response (complete and partial) rate

SECONDARY OUTCOMES:
Progression-free survival
Overall survival
Tolerance
Resectability rate
Biomarkers predictive of efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Borg, PhD — Hopital Jean Minjoz
Locations (1):
- Centre Hospitalier Regional de Besancon - Hopital Jean Minjoz, Besançon, France

REFERENCES:
- [Derived] Jary M, Lecomte T, Bouche O, Kim S, Dobi E, Queiroz L, Ghiringhelli F, Etienne H, Leger J, Godet Y, Balland J, Lakkis Z, Adotevi O, Bonnetain F, Borg C, Vernerey D. Prognostic value of baseline seric Syndecan-1 in initially unresectable metastatic colorectal cancer patients: a simple biological score. Int J Cancer. 2016 Nov 15;139(10):2325-35. doi: 10.1002/ijc.30367. Epub 2016 Aug 13. PMID 27472156